CLINICAL TRIAL: NCT02111473
Title: Phase 4 Study of Effect of Testosteron Replacement Treatment on the Fibroblast Growth Factor-23, Asymmetric Dimethylarginine and Vitamin D Levels in the Congenital Hypogonadotropic Hypogonadism
Brief Title: The Effect of Testosteron Replacement Treatment on the Fibroblast Growth Factor-23, Asymmetric Dimethylarginine and Vitamin D Levels in the Congenital Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, cem haymana, MD, Gulhane School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSM-032014
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Hypogonadism
Keywords: endothelial dysfunction; bone mineral metabolism; testosteron replacement treatment
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- testosterone (Other): testosterone 250 mg injection per 3-4 weeks for 6 months
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone 250 mg injection per 3-4 weeks for 6 months
  Other Names: sustanon 250 mg

SUMMARY:
The study is designed to answer the following questions:

1) What is the effect of testosteron replacement treatment on the endothelial dysfunction.

2/ What is the effect of testosteron replacement on the bone mineral metabolism.

DETAILED DESCRIPTION:
this is an interventional study which is examine the effect of testosteron replacement treatment on the endothelial dysfunction and bone mineral metabolism in hypogonadotropic hypogonadal patients.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Congenital hypogonadism
* Treatment Naive

Exclusion Criteria:

* Previous history of androgen replacement
* Hypertension
* Diabetes mellitus

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the effect of testosteron replacement treatment on the Fibroblast Growth Factor-23. | 6 months
  Plasma FGF-23 levels were determined by ELISA, (Human Intact FGF-23 ELISA Kit, Inc., San Clement, CA, USA).
the effect of testosteron replacement treatment on the asymmetric dimethylarginine. | 6 months
  Plasma ADMA levels were determined by ELISA (Immunodiagnostic, Bernheim, Germany)
the effect of testosteron replacement treatment on the vitamin D levels. | 6 months.
  Plasma 25-OH vitamin D3 levels were measured by Immuchrom kits (Hessen, Germany) using isocratic HPLC method with UV detector in Prominence HPLC system.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)